CLINICAL TRIAL: NCT04890418
Title: Risk Factors and Prevention of Severe Pain Upon Cessation of a Peripheral Nerve Block. A Prospective Randomized Study in Ambulatory Patients Undergoing Upper Limb Bone Surgery Under Single Shot Axillary Plexus Block
Brief Title: Risk Factors and Prevention of Severe Pain Upon Cessation of a Peripheral Nerve Block
Acronym: PRPK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/05JUL/303
Record Dates: First submitted 2020-03-03; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Surgery
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The local pharmacy department is in charge of unmasking the drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study drug (Active Comparator): 0.3 mg/kg intravenous ketamine diluted into 10mL saline after the realization of peripheral nerve block (PNB), before tourniquet set up and beginning of surgery
  Interventions: Drug: Ketalar, 5 mg/mL Injectable Solution
- Placebo (Placebo Comparator): 10 mL 0.9% saline after the realization of PNB, before tourniquet set up and beginning of surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketalar, 5 mg/mL Injectable Solution — The patients will receive (slow intravenous injection) 0.3 mg/kg intravenous ketamine diluted by the pharmacy department into 10mL saline after the realization of PNB but before tourniquet set up and before start of surgery.
  Other Names: Active comparator
  Arms: Study drug
Other: Placebo — The patients will receive 10 mL of 0.9% saline. This injection is also performed after the realization of PNB but before tourniquet set up and before start of surgery.
  Other Names: Placebo comparator
  Arms: Placebo

SUMMARY:
Risk factors and Prevention of severe Pain upon cessation of a peripheral nerve block. A prospective randomized study in ambulatory patients undergoing upper limb bone surgery under single shot axillary plexus block.

DETAILED DESCRIPTION:
Pain in the course of upper limb bone surgery is a major source of discomfort for patients during postoperative time.

Severe post-operative pain is a risk factor for chronic pain. Use of a well-known molecule, regularly used in anesthesiology. Prospective double-blind study on 120 patients. Pain rebound upon awakening of the axillary plexus during upper limb bone surgery is a frequent phenomenon in post-operative follow-up of patients.

The anti-hyperalgesic properties of ketamine could be a benefit against this effect.

No studies have combined intravenous ketamine with localoregional anesthesia to reduce pain upon its release.

This may improve patients' post-operative comfort. The patients will be randomized in 2 groups and allocated to receive (slow intravenous injection) either 0.3 mg/kg intravenous ketamine diluted into 10mL saline or 10 mL 0.9% saline after the realization of PNB, before tourniquet set up and beginning of surgery.

ELIGIBILITY:
Inclusion Criteria:

* any ambulatory upper limb bone surgery carried out under axillary PNB

Exclusion Criteria:

* Refusal to participate
* Contraindication to the use of ketamine
* Contraindication to regular use of postoperative analgesics like non-steroidal anti-inflammatory drugs and paracetamol
* Pregnant woman
* Diabetic patient
* Vascular patient
* Cognitive disorders
* Inability to answer perioperative questionnaires (language problem)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
incidence of severe postoperative rebound pain | from surgery to 30 days post operation
  Rebound pain after PNB is defined as a Numerical rating Scale of 7 or more.

SECONDARY OUTCOMES:
To measure the impact of ketamine on the level of "rebound pain" in patients with central sensitivity using the Numerical Rating Scale | from surgery to 30 days postoperatively
  Central sensitivity analyzed by a questionnaire and by Numerical Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided